CLINICAL TRIAL: NCT03754166
Title: Feasibility of Modified Constraint-induced Movement Therapy Combined With Visual-spatial Cueing Strategy in Patients With Acute Stroke
Brief Title: Feasibility of Constraint-induced Therapy Combined With Visual-spatial Cueing Strategy in Patients With Acute Stroke
Acronym: ITHEMICAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study non feasible following changes in organisation of service
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC18_0288
Record Dates: First submitted 2018-11-20; First posted 2018-11-27 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constraint-induced movement therapy (Experimental): Patient's unaffected arm is restrained, by a glove including thumb, during activities of daily life (bathing, grooming, dressing and feeding = approx. 4h/day).
  Visual spatial cueing is displayed in the bedroom and the bathroom.
  Interventions: Other: Constraint-induced movement therapy
- Usual care (No Intervention): Usual care of the neurovascular unit. = No constraint, no cueing, and same physiotherapy intervention as experimental arm.

INTERVENTIONS:
Other: Constraint-induced movement therapy — Patient's unaffected arm is restrained, by a glove including thumb, during activities of daily life (bathing, grooming, dressing and feeding = approx. 4h/day).
  Visual spatial cueing is displayed in the bedroom and the bathroom.
  Other Names: Visual-spatial cueing : top down
  Arms: Constraint-induced movement therapy

SUMMARY:
The aim of this study is to test the feasibility of a constraint intervention combined with visual-spatial cueing strategy in patients with acute stroke to improve their daily life activities.

DETAILED DESCRIPTION:
As part of treatment in acute stroke (from D0 to D14), the investigators were able to observe that despite motor recovery during physiotherapy sessions, it remained difficult for some patients to use their affected arm (AA) during activities of daily life (ADL). This mechanism of "learned non-use" would be due to a cognitive process decreasing the use of the AA and could partly explain that 75% of patients maintain an upper limb deficit at 3-6 month post-stroke.

In order to combat this phenomenon, a bottom up method (sensorimotor action on the deficit) of constraint-induced movement therapy (CIMT) has been developed and consists in immobilizing the unaffected arm to force the use of the AA.

This technique has proved its effectiveness in the chronic phase and has also recently been proven to improve motor performance in the acute phase. Transposing progress on ADL, however, remains difficult because CIMT does not contain adequate behavioral strategies.

To help the patient mobilize these strategies, coupling of CIMT with a top-down method (conscious action on motor skills) has been successfully tested as an intervention of an occupational therapist with the patient at least 1h / day. This intervention remains not compatible with the investigators care organization because the caregiver can not spend that amount of time with each patient.

Investigators therefore propose to associate CIMT with another top down technique: visual-spatial cueing (use of panels and/or visual messages to encourage the conscious use of the AA) and investigators want to evaluate the effectiveness of this treatment on learning transfer to ADL.

The objective of our study will be to test the feasibility of setting up such an intervention.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient in neurovascular unit for stroke
* Time since stroke between 2 and 4 days
* Movement capacity of the upper arm (against gravity) :
* Ability to extend actively the metacarpophalangeal and interphalangeal joints at least 10°, and the wrist 20°
* Ability to bend actively the elbow at least 45°
* Ability to bend and abduct actively the shoulder at least ≥ 45°
* Age ≥ 18 years old
* Patient agreement to join the study
* Patient covered by french social security

Exclusion Criteria:

* Excessive spasticity : score > 2 on the modified Ashworth scale
* Excessive pain in the affected arm : score ≥ 4 on the visual analogue scale
* Joint limitation on the affected arm
* Patient under guardianship or curatorship
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Number of tasks realized per protocol between the two arms | Day 15
  Variances to a predetermined checklist

SECONDARY OUTCOMES:
Arm motor function | Day 0, Day 15 and Month 3
  Action Research Arm Test
Pain evolution | Day 0, Day 7, Day 15 and Month 3
  Use of Visual analogue scale to determine the degree of pain on a scale from 0 to 10 (0: meaning no pain, 10 being maximal tolerable pain)
Anxiety and Depression evolution | Day 0, Day 7, Day 15 and Month 3
  Use of Hospital Anxiety and Depression Scale. This scale has 14 items in total, 7 items for Anxiety and 7 for Depression. Each item is rated from 0 to 3. score of 0 meaning normal, score 3 meaning abnormal.
Situation of patient after neurovascular unit | Month 3
  Indication of patient 's situation at the end of the study: either Rehabilitation center, Nursing homes, Home or Other

CONTACTS AND LOCATIONS:
Overall Officials: Ambre Komonski, Principal Investigator — Nantes University Hospital
Locations (1):
- Service de Neurologie, CHU Nantes, Nantes, France